CLINICAL TRIAL: NCT00890422
Title: Clinical Study to Test the Immunogenicity of Variant Schedules for TBE Rapid Immunisation Using Inactivated TBE (FSME) Vaccine
Brief Title: Evaluation of Immunogenicity of Different Tick Borne Encephalitis (TBE) Fast Protective Traveler Schemes With Inactivated TBE Whole Virus Vaccine
Acronym: immunisation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Elisabethinen Hospital (Other)
Collaborators: Baxter Healthcare Corporation (Industry); ASOKLIF (Unknown)
Responsible Party: Helmut Mittermayer/Univ.Prof. Dr., Elisabethinen Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: ASOKLIF 0608/MI; Eudract number: 2006-006955-10
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Tick Borne Encephalitis
Keywords: encephalitis; FSME; central european encephalitis
MeSH Terms: conditions — Encephalitis, Tick-Borne; Encephalitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1FSME vaccination (Experimental): 2 vaccination on day 0
  Interventions: Biological: FSME vaccination (FSME-Immun)
- 2 FSME vaccination (Experimental): 1 vaccination on day 0 and one vaccination on day 4
  Interventions: Biological: FSME vaccination (FSME-Immun)
- 3 FSME vaccination (Experimental): 2 vaccinations on day 0 and 1 vaccination on day 4
  Interventions: Biological: FSME vaccination (FSME-Immun)

INTERVENTIONS:
Biological: FSME vaccination (FSME-Immun) — intra muscular 0.5 ml
  Other Names: FSME-Immun 0.5 ml

SUMMARY:
The study aims to answer this question: whether adequate immunity can be achieved in a short time, that is, by a rapid immunisation process, using at least one of 3 new TBE immunisation schedules? The investigators will test the immunogenicity (the degree of immunity achieved) of each of the immunisation schedules at various times after the injections. If the results of this clinical study are positive, it may then be possible to develop the most successful immunisation schedule so that it can be used routinely. This means that the results of the clinical study have an enormous practical value in preventing TBE in people travelling or moving into areas with a high TBE risk.

DETAILED DESCRIPTION:
The data from at least 99 individuals will be needed if the study is to draw reliable conclusions. One-third of these individuals will receive 3 injections in all: 2 on the first day and the third injection 4 days later (immunisation schedule 1). Another one-third will receive 2 injections in all: one on the first day and one injection 4 days later (immunisation schedule 2). The remaining one-third will also receive 2 injections, both of these on the first day (immunisation schedule 3). Participants will be assigned completely randomly (by chance) to one of these three groups. So each participant stands a 33% chance (a 1:2 chance) of receiving any one particular immunisation schedule. If you agree to take part, the process will be as follows:

Brief Overview of the Course of the Clinical Study:

Vaccination scheme 1

Vaccination scheme 2

Vaccination scheme 3

Vaccinations:

I = Vaccination with FSME-IMMUN 0,5ml

* Scheme 1: 2 vaccinations at U1 (day 0), one injection into the left and the right upper arm each, 1 vaccination at U2 (day 4), injection into the left upper arm
* Scheme 2: one vaccination at U1 (day 0) and at U2 (day 4), injections into the left upper arm each
* Scheme 3: 2 vaccinations at U1 (day 0), one injection into the left and the right upper arm each

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* FSME antibody level < 7IU/ml (ELISA), retrospective
* FSME antibody (IgG) < 63 VIEU/ml (ELISA), retrospective
* FSME antibody (IgM) negative
* FSME antibody inhibition capacity <1:10-retrospective
* available for the next 56 days

Exclusion Criteria:

* age not 19 or over 65
* pregnancy
* risk of becoming pregnant

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-11 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
achievement of FSME-Antibody-level (IgG) >25IU/ml at visit U2, U3, U4, U5, U6, U7, U8 and U9-yes/no achievement of FSME antibody-level (IgG) of >126VIEU/ml at U2, U3;U4, U5, U6, U7, U8 and U9-yes/no | U2 (=day4) U3 (=day7) U4 (=day10) U5 (=day 14) U6 (=day21) U7 (=day28) U8 (=day42) U9 (=day56)

SECONDARY OUTCOMES:
FSME antibody level at U2, U3, U4, U5, U6, U7, U8 and U9 | U2 (=day4) U3 (=day7) U4 (=day10) U5 (=day 14) U6 (=day21) U7 (=day28) U8 (=day42) U9 (=day56)

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Mittermayer, Principal Investigator — Elisabethinen Hospital
Locations (2):
- Elisabethinen Hospital, Linz, Upper Austria, Austria
- nemocnice ceske Budejovice, České Budějovice, Czechia

REFERENCES:
- See also: ethics committee of the Elisabethinen hospital — http://www.elisabethinen.or.at